CLINICAL TRIAL: NCT02880228
Title: Phase 2 Trial of Pembrolizumab, Lenalidomide, and Dexamethasone for Initial Therapy of Newly Diagnosed Multiple Myeloma Eligible for Stem Cell Transplantation
Brief Title: Pembrolizumab, Lenalidomide, and Dexamethasone in Treating Patients With Newly Diagnosed Multiple Myeloma Eligible for Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1588; NCI-2016-01290 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1588 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-04

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lenalidomide, dexamethasone, pembrolizumab) (Experimental): Patients receive lenalidomide PO daily on days 1-21 and dexamethasone PO daily on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV over 30 minutes on days 1 and 22 of course 1, day 15 of course 2, and day 8 of course 3. Courses 1-3 repeat beyond 3 courses in the absence of disease progression or unacceptable toxicity. Patients may undergo stem cell transplantation after 4 courses of treatment.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab, lenalidomide, and dexamethasone work in treating patients with newly diagnosed multiple myeloma that are eligible for stem cell transplant. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab, lenalidomide, and dexamethasone may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the very good partial response (VGPR) or better response rate (>= VGPR) after 4 cycles of pembrolizumab added to standard doses of lenalidomide and dexamethasone, when used as initial therapy in patients with previously untreated symptomatic multiple myeloma (MM) in patients, who are considered eligible for stem cell transplantation.

SECONDARY OBJECTIVES:

I. To determine the >= partial response (PR) rate after 4 cycles of treatment with pembrolizumab added to standard doses of lenalidomide and dexamethasone.

II. To determine the >= VGPR response rate at any time during treatment with pembrolizumab added to standard doses of lenalidomide and dexamethasone.

III. To determine the progression free survival and overall survival among patients with previously untreated symptomatic MM following treatment with the combination of pembrolizumab, lenalidomide and dexamethasone.

IV. To determine the toxicities associated with pembrolizumab added to standard doses of lenalidomide and dexamethasone in patients with previously untreated symptomatic MM.

V. To determine the success rate of stem cell collection following initial therapy with the combination of pembrolizumab, lenalidomide and dexamethasone in patients with newly diagnosed MM.

TERTIARY OBJECTIVES:

I. PDL-1 expression on myeloma cells and non-tumor cell compartments from the bone marrow will be assessed at baseline.

II. Measures of T-cell activation / exhaustion will be assessed at baseline and after cycle 1, cycle 2, cycle 3, and cycle 4.

III. Natural killer (NK) cell function and numbers will be evaluated at baseline and after cycle 1, cycle 2, cycle 3, and cycle 4.

OUTLINE:

Patients receive lenalidomide orally (PO) daily on days 1-21 and dexamethasone PO daily on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab intravenously (IV) over 30 minutes on days 1 and 22 of course 1, day 15 of course 2, and day 8 of course 3. Courses 1-3 repeat beyond 3 courses in the absence of disease progression or unacceptable toxicity. Patients may undergo stem cell transplantation after 4 courses of treatment.

After completion of study treatment, patients are followed up every 3 months or 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis and previously untreated active multiple myeloma by International Myeloma Working Group (IMWG) diagnostic criteria for multiple myeloma
* Calculated creatinine clearance (using Cockcroft-Gault equation) >= 30 mL/min
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelet count >= 75000/mm^3
* Hemoglobin >= 8.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN
* Prior therapy for the treatment of solitary plasmacytoma is permitted, but > 7 days should have elapsed from the last day of radiation

  * NOTE: Prior therapy with clarithromycin, dehydroepiandrosterone (DHEA), anakinra, pamidronate, or zoledronic acid is permitted; any additional agents not listed must be approved by the principal investigator
* Measurable disease of multiple myeloma as defined by at least ONE of the following:

  * Serum monoclonal protein >= 1.0 g/dL
  * > 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Provide written informed consent
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Willing to follow strict birth control measures as suggested by the study

  * Female patients: If they are of childbearing potential, must agree to one of the following:

    * Practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
  * Male patients: even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 120 days after the last dose of study drug, OR
    * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide consent to Institutional Review Board (IRB) number (#) 521-93 and provide research tissue and blood specimens

Exclusion Criteria:

* Monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma
* Prior cytotoxic chemotherapy or corticosteroids for the treatment of multiple myeloma

  * NOTE: Prior corticosteroid use for the treatment of non-malignant disorders is permitted
* Diagnosed or treated for another malignancy =< 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease.

  * NOTE: Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other co-morbidity which would interfere with patient's ability to participate in trial, e.g. uncontrolled infection, uncompensated heart or lung disease
* Other concurrent chemotherapy or any ancillary therapy considered investigational

  * NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Peripheral neuropathy >= grade 3 on clinical examination or grade 2 with pain during the screening period
* Major surgery =< 14 days prior to study registration
* Radiotherapy =< 14 days prior to registration

  * NOTE: If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of study drugs
* Participation in any other clinical trials with other investigational agents not included in this trial, =< 21 days prior to registration
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs)

  * NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Active infection requiring systemic therapy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Received a live vaccine =< 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2018-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Lenalidomide, Dexamethasone, Pembrolizumab): Patients receive 25 mg lenalidomide PO daily on days 1-21 and 40 mg dexamethasone PO daily on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also receive 200 mg pembrolizumab IV over 30 minutes on days 1 and 22 of course 1, day 15 of course 2, and day 8 of course 3. Courses 1-3 repeat beyond 3 courses in the absence of disease progression or unacceptable toxicity. Patients may undergo stem cell transplantation after 4 courses of treatment.
Period: Overall Study
Arm/Group | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients that began protocol treatment are included in this analysis.
Arm/Group | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab)
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 59 [42 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Complete Response Plus Very Good Partial Response (VGPR)
Description: The International Myeloma Working Group response criteria was used to assess response to therapy. The proportion of VGPR response at any time during treatment with pembrolizumab added to lenalidomide and dexamethasone will be estimated by the number of patients achieving a VGPR, CR, or sCR at any time divided by the total number of evaluable patients. A very good partial response (VGPR) is defined as as a demonstration of:
  * Serum and urine M-component detectable by immunofixation but not on electrophoresis c or
  * greater than 90% reduction in serum m-component and urine m-component <100 mg/24 h
  * If the only measurable disease is FLC, a ≥90% reduction in the difference between involved and involved FLC levels
  The proportion of successes will be estimated by the number of patients demonstrating a VGPR or better divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: Up to 112 days
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab)
Number analyzed (Participants) | 11
proportion of participants | 0 [0 to 0.28]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from registration to the earliest date of documentation of disease progression or death due to any cause. Patients who receive subsequent treatment for myeloma before disease progression will be censored on the date of their last disease assessment prior to initiation of the subsequent treatment. Transplant will not be considered subsequent treatment. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 3 years
Population: All patients that began protocol treatment were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab)
Number analyzed (Participants) | 11
months | NA [NA to NA] — Too few events occurred to estimate the median and confidence interval.

3. Secondary Outcome: Partial Response (PR)
Description: The PR response after 4 cycles of induction treatment with pembrolizumab added to lenalidomide and dexamethasone will be estimated by the number of patients who achieve a PR, VGPR, CR, or sCR after 4 cycles divided by the total number of evaluable patients. A PR is defined by the following criteria:>
  * If present at baseline, ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein or to <200 mg/24hrs>
  * If the only measurable disease is FLC, a ≥50% reduction in the difference between involved and involved FLC levels>
  * If the only measurable disease is BM, a ≥50% reduction in BM PC's (provided the baseline PC's was ≥30%)>
  * If present at baseline, ≥50% reduction in the size of soft tissue plasmacytomas>
  Exact binomial 95% confidence intervals for the true success rate will be calculated.
Time Frame: Up to 112 days
Population: Only patients that completed 4 cycles of treatment were included in this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab)
Number analyzed (Participants) | 5
proportion of participants | 0 [0 to 0.52]

4. Secondary Outcome: Proportion of Successful Stem Cell Collection
Description: The proportion of successful stem cell collection following initial therapy with the combination of pembrolizumab, lenalidomide and dexamethasone in patients with newly diagnosed MM will be estimated by the number of patients with a successful stem cell collection divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true successful proportion will be calculated.
Time Frame: Up to 112 days
Population: Only patients that completed 4 cycles of treatment were eligible for this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab)
Number analyzed (Participants) | 5
proportion of participants | 0.4 [0.05 to 0.85]

5. Secondary Outcome: Survival Time
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From time of registration to death due to any cause, assessed up to 3 years
Population: All patients that began protocol treatment are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab)
Number analyzed (Participants) | 11
months | NA [NA to NA] — Too few events occurred to estimate a median and confidence interval.

ADVERSE EVENTS:
Time Frame: Adverse events were collected after every 28 day cycles during treatment, up to 7 cycles.
Arm/Group | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab) (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Lenalidomide, Dexamethasone, Pembrolizumab) (N=11)
Anemia (Blood and lymphatic system disorders) | 9 (25)
Constipation (Gastrointestinal disorders) | 4 (13)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 9 (27)
Creatinine increased (Investigations) | 2 (2)
Hemoglobin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 5 (9)
White blood cell decreased (Investigations) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02880228/Prot_SAP_000.pdf